CLINICAL TRIAL: NCT06646406
Title: Evaluation of a Multilevel Intervention on Adult COVID-19 and Influenza Vaccination Rate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: ModernaTX, Inc. (Industry)
Responsible Party: Principal Investigator, Lila J. Rutten, Professor of Health Services Research; Chair, Division of Epidemiology, Department of Quantitative Health Sciences, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 24-007738
Record Dates: First submitted 2024-09-30; First posted 2024-10-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: COVID-19 Immunisation; Influenza Vaccine
Keywords: Adult; Vaccination; Influenza vaccines; COVID-19 Vaccines; Primary Health Care; Reminder Systems; Clinician communication; Patient communication
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient letter and clinician communication (Experimental): Each patient will be mailed a letter and each patient's clinician will receive a monthly email communicating information about making a strong recommendation for influenza and COVID-19 vaccination
  Interventions: Behavioral: Patient letter and clinician communication
- No intervention (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Patient letter and clinician communication — Single mailing to patients from practice with a reminder that the influenza and COVID-19 vaccines are due, and monthly emailing to the patients' clinicians with information about how to make a strong recommendation for those vaccines
  Other Names: Reminder systems; Clinician communication
  Arms: Patient letter and clinician communication

SUMMARY:
The study will test two tactics to improve uptake of two vaccines in adults. The vaccines prevent COVID-19 and influenza. Both are common and harmful. Most adults do not get either vaccine. This is despite strong recommendations that all adults get both vaccines.

The study will involve adult patients at eight Mayo Clinic primary care practices in Rochester and Kasson. The study will test the two tactics together. Four clinics will get the two tactics. The other four clinics will not. The study will randomly assign the two tactics to the clinics. One tactic is to send a letter by US mail to the patient. The letter will state strong recommendations on getting both vaccines now. It will tell patients how to get the vaccines now. The second tactic is to send monthly emails to clinicians. It will remind them to use every visit to vaccinate patients against COVID-19 and influenza. The study will compare the uptake of the two vaccines after six months in the clinics with and without the two tactics.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 years and older
* Patients empaneled to 1 of 8 adult primary care practices as of September 2024

Exclusion Criteria:

* Patients 18 years or younger
* Patients not empaneled to 1 of 8 adult primary care practices as of September 2024

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114165 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 vaccine uptake | 7.5 months
  Rates of at least one dose of single licensed 2024-2025 COVID-19 vaccine among adult patients at eight Mayo Clinic primary care practices
Influenza vaccine uptake | 9 months
  Rates of at least one dose of single licensed 2024-2025 trivalent influenza vaccine among adult patients at eight Mayo Clinic primary care practices

CONTACTS AND LOCATIONS:
Overall Officials: Lila J. Rutten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States